CLINICAL TRIAL: NCT07312838
Title: Ultrasound Evaluation of Fetal Liver Length and Volume as Novel Markers of Glycemic Impact in Pregnancy: A Prospective Cohort Study
Brief Title: Evaluation of Glycemic Impact on Fetal Liver Length and Volume by Ultrasound in Pregnancy
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yousef Ahmed Mahmoud Ahmed, Dr. Yousef Ahmed Mahmoud Ahmed, Assiut University
Other Study IDs: Fetal liver parameters by U/S
Record Dates: First submitted 2025-11-24; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Gestatiaonl Diabetes Mellitus; FETAL LİVER VOLUME
Keywords: Ultrasound; Fetal liver length; Fetal liver volume; Gestational diabetes mellitus
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary aim of this study is to evaluate whether fetal liver length and volume, as assessed by ultrasound, can serve as reliable markers of the metabolic impact of Gestational Diabetes Mellitus (GDM) on the fetus.

DETAILED DESCRIPTION:
Maternal hyperglycemia during pregnancy, even at levels below the diagnostic threshold for gestational diabetes mellitus (GDM), is associated with adverse outcomes such as macrosomia, neonatal hypoglycemia, and long-term metabolic risk in offspring. Current clinical assessment of glycemic impact relies primarily on maternal glucose testing, such as the oral glucose tolerance test (OGTT), and indirect fetal anthropometric markers including abdominal circumference or estimated fetal weight . However, these measures may not fully reflect the fetal metabolic response to maternal hyperglycemia . Emerging evidence suggests that the fetal liver is highly sensitive to maternal glycemic status due to its central role in glucose uptake, glycogen storage, and lipid metabolism . Ultrasound studies have demonstrated that fetuses of mothers with GDM often show increased liver length and volume compared with normoglycemic controls, and these changes can occur before overt increases in overall fetal size .Thus, fetal liver measurements may provide an earlier and more direct marker of intrauterine glycemic exposure . Currently, the strategy for evaluating glycemic impact in pregnancy is based on maternal glucose testing and late-gestation fetal growth assessment, which may delay timely intervention . Moreover, there is no widely accepted ultrasound marker that specifically reflects fetal metabolic adaptation to hyperglycemia . The rationale of this research is to evaluate fetal liver length and volume by ultrasound as novel markers of glycemic impact in pregnancy. By establishing their relationship with maternal glycemic status, this study aims to determine whether fetal liver measurements can serve as an early, non-invasive, and practical tool to identify at-risk pregnancies, thereby paving the way for improved monitoring and timely intervention.

ELIGIBILITY:
Inclusion Criteria:

1. gestational age 24wks-36wks by an early pregnancy ultrasound exam including CRL length
2. normal maternal blood sugar levels in early pregnancy
3. diagnosed as GDM
4. singleton viable pregnancy
5. agree to include in study

Exclusion Criteria:

1. preexisting diabetes
2. fetal congenital anomalies or chromosomal abnormalities
3. maternal chronic illnesses (e.g. Hypertension , thyroid disorders)
4. multiple pregnancies

Ages: 18 Years to 52 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: Deep learning machine
  This prospective cohort consisted of pregnant women recruited from the antenatal clinics and fetal-medicine unit at Women's Health Hospital at Assiut University , between [December 2025 - March 2029]. Participants were enrolled at the time of their routine mid-trimester/anomaly ultrasound (targeted recruitment window 24weeks gestation for mid-trimester measures, with repeat/late scans at 36 weeks when required for longitudinal liver volume assessment)
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-03-28 (Estimated); Study Completion 2028-03-28 (Estimated)

PRIMARY OUTCOMES:
Correlation of fetal liver length with maternal glycemic state | 12 weeks
  Correlation of fetal liver length with maternal glycemic state
Comparison of fetal liver length | 12 weeks
  Comparison of fetal liver length between women with gestational diabetes mellitus (GDM) and normoglycemic pregnancies.
Correlation of fetal liver volume with maternal glycemic state | 12 weeks
  Correlation of fetal liver volume with maternal glycemic state
Comparison of fetal liver volume between women with gestational diabetes mellitus (GDM) and normoglycemic pregnancies. | 12 weeks
  Comparison of fetal liver volume between women with gestational diabetes mellitus (GDM) and normoglycemic pregnancies.

SECONDARY OUTCOMES:
Correlation of fetal liver size with standard fetal biometry | 12 weeks
  Correlation of fetal liver size with standard fetal biometry (abdominal circumference, estimated fetal weight).
Relationship of fetal liver measurements with neonatal outcomes | 12 weeks
  Relationship of fetal liver measurements with neonatal outcomes (birth weight, macrosomia, neonatal hypoglycemia
Comparison of abdominal circumference with fetal liver volume | 12 weeks
  Comparison of abdominal circumference with fetal liver volume
Comparison of abdominal circumference with fetal liver length | 12 weeks
  Comparison of abdominal circumference with fetal liver length

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/27603367/
- See also: Related Info — https://journals.lww.com/mfm/fulltext/2019/10000/role_of_ultrasonography_in_pregnancies_complicated.6.aspx
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC8346004/